CLINICAL TRIAL: NCT00112008
Title: A Multi-Center, Single-Arm Study Evaluating De Novo Once Every Two Week Darbepoetin Alfa Dosing in Subjects With Chronic Kidney Disease (CKD) Not Receiving Dialysis
Brief Title: Study for Subjects With Chronic Kidney Disease(CKD) Not Receiving Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030237
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Kidney Disease; Kidney Disease
Keywords: Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Anemia

ARMS (1):
- darbepoetin alfa (Experimental)
  Interventions: Drug: De Novo Administration of Darbepoetin Alfa

INTERVENTIONS:
Drug: De Novo Administration of Darbepoetin Alfa — Administration Q2W for 18 weeks. starting dose is 0.75 mcg/kg rounded to the nearest dose: 20, 30, 40, 50, 60, 80, 100, 150, 200 0r 300 mcg. Titrate to maintain Hb within 11.0 - 13.0 g/dL

SUMMARY:
The proposed study is designed to test a novel dosing paradigm that would facilitate the treatment of anemia in CKD patients not on dialysis. Anemic patients who are not currently receiving ESA therapy will be dosed with darbepoetin alfa Q2W for 18 weeks.

ELIGIBILITY:
Inclusion Criteria: - Diagnosis of CKD and not expected to initiate dialysis for the duration of the study - Estimated glomerular filtration rate (eGFR): greater than or equal to 15 mL/min and less than or equal to 60 mL/min measured by the following modified MDRD (Modification of Diet in Renal Disease) equation: eGFR = 186 x [serum creatinine]-1.154 x [Age]-0.203 x [0.742 if subject is female] x [1.212 if subject is black] - Clinically stable, in the judgment of the investigator - Mean Hb greater than or equal to 11.0 g/dL to less than or equal to 13.0 g/dL (mean of 2 values drawn at least 3 days apart during the screening period) - Transferrin saturation (Tsat) greater than or equal to 15.0% - Serum vitamin B12 and folate levels above the lower limit of the normal range - Receiving stable Q2W subcutaneous (SC) doses of Aranesp® (darbepoetin alfa). A stable dose is defined as less than or equal to a 25% change in dose over the 6-week period immediately prior to enrollment and with no missed doses in this period Exclusion Criteria: - Prior recipient or scheduled to receive a kidney transplant - Diastolic blood pressure (BP) greater than 110 mm Hg or systolic BP greater than 180 mm Hg during screening - Acute myocardial ischemia - Hospitalization for congestive heart failure or myocardial infarction within 12 weeks before enrollment - Parathyroid hormone level greater than 1500 pg/mL - Major surgery within 12 weeks before enrollment (excluding vascular access surgery) - Currently receiving antibiotic therapy for systemic infection - Known positive HIV antibody or positive hepatitis B surface antigen - Clinical evidence of current malignancy and/or receiving systemic chemotherapy/radiotherapy with the exception of basal cell or squamous cell carcinoma of the skin and cervical intraepithelial neoplasia - Red blood cell (RBC) transfusions within 8 weeks before enrollment - Androgen therapy within 8 weeks before enrollment - Systemic hematologic disease (e.g., sickle cell anemia, myelodysplastic syndromes, hematologic malignancy, myeloma, hemolytic anemia) - Any disorder that may impact (in the judgment of the investigator) the ability to give informed consent for participation in this study - Pregnant or breast-feeding women - All subjects must practice adequate contraception (in the judgment of the investigator) throughout this trial - Treatment with an investigational agent or device within 30 days before enrollment or scheduled to receive an investigational agent other than those specified by this protocol during the course of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-05; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects achieving a Hb ≥ 11.0 g/dL | Entire Study

SECONDARY OUTCOMES:
Hb values over the duration of the study | Entire Study
Darbepoetin alfa doses over the duration of the study | Entire Study
Frequency, severity, and relationship to treatment for adverse events and changes in laboratory parameters and blood pressure | Entire Study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Silver MR, Geronemus R, Krause M, Chen CY, Kewalramani R, Stehman-Breen C. Anemia treatment with Q2W darbepoetin alfa in patients with chronic kidney disease naive to erythropoiesis-stimulating agents. Curr Med Res Opin. 2009 Jan;25(1):123-31. doi: 10.1185/03007990802594818. PMID 19210145
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20030237.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/